CLINICAL TRIAL: NCT00486291
Title: A Phase 2, Randomized, Double Blind, Parallel Design Study Comparing the Efficacy and Safety of VI-0521 to Placebo in the Glycemic Management of Obese Diabetic Adults
Brief Title: Study of VI-0521 Compared to Placebo in the Glycemic Management of Obese Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OB-202
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes, Obese diabetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Phentermine 15mg/topiramate 100mg
  Interventions: Drug: VI-0521
- 2 (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VI-0521 — phentermine 15mg/topiramate 100mg
  Arms: 1
Drug: Placebo — matched placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VI-0521 compared to placebo in the glycemic management of obese diabetic adults.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Type 2 Diabetes
* BMI 27-42
* Specified diet/exercise and/or diabetes medications

Exclusion Criteria:

* BP > 150/95
* Stroke/MI/unstable cardiovascular disease within 6 months
* Clinically significant renal, hepatic, or psychiatric disease
* Unstable thyroid disease or replacement therapy
* Nephrolithiasis
* Obesity of known genetic or endocrine origin
* Participation in a formal weight loss program or lifestyle intervention
* History of glaucoma
* Pregnancy or breastfeeding
* Alcohol abuse
* Eating disorder
* Excluded medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Troupin, MD, MBA, Study Director — VIVUS LLC
Locations (9):
- United States (9):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Spring Valley, California
  - Research Site, Walnut Creek, California
  - Research Site, Bethesda, Maryland
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred in 10 investigative sites in the U.S. between May 2007 and July 2007
Groups:
- Active: Phentermine 15mg/topiramate 100mg
Period: Overall Study
Arm/Group | Active | Placebo
Started | 105 (3 subjects discontinued prior to first dose) | 105 (1 subject discontinued prior to first dose)
Completed | 89 | 76
Not Completed | 16 | 29
Not completed — Adverse Event | 3 | 4
Not completed — Lost to Follow-up | 3 | 7
Not completed — protocol non-compliance | 10 | 15
Not completed — requirement for restricted medication | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 102 | 104 | 206
Age Continuous [Mean (Standard Deviation); unit: years] | 50.2 (8.39) | 48.5 (9.72) | 49.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 64 | 141
  Male | 25 | 40 | 65
Region of Enrollment [Number; unit: participants]
  United States | 102 | 104 | 206

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 28.
Time Frame: Baseline to 28 weeks
Population: Intent-to-treat Last-observation-carried-forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Active: Phentermine 15mg and topiramate 100mg
Arm/Group | Active | Placebo
Number analyzed (Participants) | 99 | 101
percent change | -1.1 (0.12) | -0.6 (0.11)
Statistical Analysis 1: Comparison: Active vs Placebo; It is anticipated that the pooled standard deviation (SD) of the change from baseline in HbA1c will be between 1.0 and 1.5. With 90 subjects per treatment group the study will have 90% power (two-sided alpha=0.05) to detect a mean difference between groups of 0.486 for SD=1.0, and a mean difference between groups of 0.729 for SD=1.5; Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.9 to -0.2], Standard Error of Mean 0.16

2. Secondary Outcome: Absolute Weight Change (kg) From Baseline to Week 28
Time Frame: Baseline to 28 weeks
Population: Intent-to-treat Last-observation-carried-forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Active | Placebo
Number analyzed (Participants) | 99 | 101
kg | -7.7 (0.57) | -1.3 (0.57)
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-8.1 to -4.9], Standard Error of Mean 0.81

ADVERSE EVENTS:
Time Frame: AEs were collected from when written informed consent was provided through 28 days after the last dose of investigational product.
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 5/102 | 6/104
Other Adverse Events (participants affected / at risk) | 85/102 | 86/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=102) | Placebo (N=104)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
anemia (Blood and lymphatic system disorders) | 1 | 0
cardiac arrest (Cardiac disorders) | 0 | 1
cardiac failure congestive (Cardiac disorders) | 0 | 2
non-cardiac chest pain (General disorders) | 0 | 1
cholelithiasis (Hepatobiliary disorders) | 1 | 0
viral infection (Infections and infestations) | 1 | 0
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
thalamic infarction (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=102) | Placebo (N=104)
upper respiratory tract infection (Infections and infestations) | 13 | 19
influenza (Infections and infestations) | 8 | 3
nasopharyngitis (Infections and infestations) | 5 | 5
bronchitis (Infections and infestations) | 5 | 3
nausea (Gastrointestinal disorders) | 18 | 5
diarrhea (Gastrointestinal disorders) | 11 | 6
constipation (Gastrointestinal disorders) | 10 | 2
dry mouth (Gastrointestinal disorders) | 8 | 1
vomiting (Gastrointestinal disorders) | 5 | 4
gastroesophageal reflux disease (Gastrointestinal disorders) | 7 | 1
paresthesia (Nervous system disorders) | 18 | 0
dizziness (Nervous system disorders) | 8 | 1
headache (Nervous system disorders) | 5 | 3
hypoesthesia (Nervous system disorders) | 5 | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
fatigue (General disorders) | 5 | 3
hypoglycemia (Metabolism and nutrition disorders) | 6 | 5
hypokalemia (Metabolism and nutrition disorders) | 6 | 1
insomnia (Psychiatric disorders) | 9 | 4
anxiety (Psychiatric disorders) | 7 | 4
vision blurred (Eye disorders) | 3 | 5
hypertension (Vascular disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.